CLINICAL TRIAL: NCT04373967
Title: A Phase III,Randomized,Parallel,Open-label,Multicenter Trial to Compare the Efficacy and Safety of Liraglutide and Victoza® in Patients With Type 2 Diabetes Inadequately Controlled by Oral Metformin Alone
Brief Title: Study to Assess the Efficacy and Safety of Liraglutide in the Treatment of Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQF2451-III-01
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQZ2451+metformin hydrochloride (Experimental): TQZ2451 injection (0.6mg qd from baseline to week 1;1.2mg qd during week 2;1.8mg qd from week 3 to week 26) + metformin hydrochloride sustained-release tablets (1500-2000mg qd)
  Interventions: Drug: Metformin Hydrochloride; Drug: TQZ2451
- Victoza®+metformin hydrochloride (Active Comparator): Victoza® (0.6mg qd from baseline to week 1;1.2mg qd during week 2;1.8mg qd from week 3 to week 26) + metformin hydrochloride sustained-release tablets (1500-2000mg qd)
  Interventions: Drug: Victoza®.; Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Victoza®. — Patients will receive Victoza®. Both products will be provided as pen-injector.
  Arms: Victoza®+metformin hydrochloride
Drug: Metformin Hydrochloride — Patients who were receiving metformin prior to study will continue to receive it during the study.
Drug: TQZ2451 — Patients will receive TQZ2451.Both products will be provided as pen-injector.
  Arms: TQZ2451+metformin hydrochloride

SUMMARY:
Liraglutide injection is a glucagon-like peptide-1 (GLP-1) analogue that activates the cyclic adenosine monophosphate (cAMP) and mitogen-activated protein kinase (MAPK) pathway by binding to the GLP-1 receptor (GLP-1R),thus,it has physiological effects such as glucose-dependent insulin synthesis and secretion, inhibition of β-cell apoptosis, promotion of β-cell proliferation and regeneration, inhibition of glucagon secretion, reduction of food intake, delay of gastric emptying, enhancement of glucose utilization in peripheral tissues and reduction of glycogen output. Liraglutide injection,developed and marketed as Victoza® by Novo Nordisk,is indicated for the treatment of patients with type 2 diabetes and was approved by the U.S. Food and Drug Administration in 2010.This 26-week trial compares the effectivity on glycaemic control,safety and immunogenicity of liraglutide injection and Victoza® in patients with type 2 diabetes inadequately controlled by oral metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as type 2 diabetes.
* Stably daily dose of metformin alone[between the dose of 1500mg and 2000mg inclusive] for at least 12 weeks prior to day of screening .
* HbA1c(glycosylated haemoglobin) of 7-11%(both inclusive).
* Body mass index (BMI) of 18.5-45 kg/m2(both inclusive).
* The patient must give informed consent to the study before the trial and voluntarily sign the informed consent form.
* The patient can communicate well with the researcher and complete the study in accordance with the research regulations.

Exclusion Criteria:

* Diagnosed as type 1 or other types of diabetes.
* Treatment with glucagon-like peptide-1 (GLP-1) receptor agonist, dipeptidyl peptidase-4 (DPP-4) inhibitor and insulin treatment within 3 months before screening.[short term (cumulative use ≤7 days) insulin therapy due to intermittent disease is excluded]
* Treatment with systemic glucocorticoid therapy within 3 months before screening[topical medication or inhaled product is excluded] .
* Treatment with Chinese medicine preparations having hypoglycemic effects within 1 month before screening.
* Patients with recurrent severe or unconscious hypoglycemia within 3 months before screening.
* Patients with acute metabolic complications (ketoacidosis, lactic acidosis or hypertonic coma, etc.) within 6 months before screening.
* History of chronic pancreatitis or idiopathic acute pancreatitis, or suffering from acute or chronic pancreatitis during screening, or blood amylase ≥ 3 times of the upper limit of normal value, or triglycerides ≥ 8.0 mmol / L.
* Fasting blood-glucose(FBG)≥15.0 mmol / L on the day of screening.
* Personal or family history of medullary thyroid carcinoma (MTC) or type 2 multiple endocrine adenoma (MEN2).
* Patients with obvious liver and kidney dysfunction (alanine aminotransferase (ALT)> 2.5 × upper normal value (ULN), aspartate aminotransferase (AST)> 2.5 ULN, glomerular filtration rate <60 Milliliter(mL) / min / 1.73m2
* Hemoglobin <lower limit of normal value.
* Hyperthyroidism is being treated or the dosage of hypothyroidism is not stable within 6 months.
* Uncontrolled or poorly treated hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg).
* Patients with decompensated heart failure (NYHA grades III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, severe arrhythmia, cardiac surgery or vascular reconstruction performed (including coronary artery bypass grafting or percutaneous coronary intervention) within 6 months before screening.
* Proliferative retinopathy or macular disease (macular edema) that requires urgent treatment.
* Malignant tumors (except basal cell carcinoma or phosphorous cell skin cancer) diagnosed within the past 5 years.
* Patients with severe chronic gastrointestinal disease (such as active peptic ulcer) and severe infections.
* People who are allergic to any of the ingredients in metformin, liraglutide injection and Victoza®.
* Participated in any other clinical trials within 3 months before screening.
* Pregnant women, lactating women and women of reproductive age who did not take appropriate contraception (sterilization, intrauterine devices, oral contraceptives or barrier contraception) during the trial.
* History of psychotropic substance abuse, alcohol abuse or drug addiction.
* Patients judged as unsuitable participants of the trial by researchers or with poor compliance.
* According to the investigators' judgment, there are seriously concomitant diseases endanger the safety of the patient or prevent the patient from completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-02 (Estimated)

PRIMARY OUTCOMES:
glycated hemoglobin (HbA1c) | week 0,week 26
  Changes in glycated hemoglobin (HbA1c) relative to baseline.

SECONDARY OUTCOMES:
Body weight | week 0,week 26
  Changes in body weight relative to baseline.
Proportion of achieving HbA1c target (<7.0% or ≤6.5%) | week 0,week 26
HbA1c change from baseline | week 0,week 14
Changes in fasting venous blood glucose (FPG). | week 0,week 14,week 26
Changes in 2h-Postprandial Blood Glucose(2h-PBG). | week 0,week 14,week 26
Changes in fasting insulin. | week 0,week 14,week 26
Changes in fasting C peptide. | week 0,week 14,week 26
Changes in systolic blood pressure. | week 0,week 14,week 26
Changes in diastolic blood pressure. | week 0,week 14,week 26
Number of adverse events and serious adverse events during exposure to trail product. | week 0-26
Number of treatment-emergent severe or blood glucose-confirmed symptomatic hypoglycaemic episodes during exposure to trail product. | week 0-26
Positive rate of liraglutide anti-drug antibody(ADA). | week 0-26
Percentage of participants with clinically significant change from baseline in vital signs. | week 0-26
Percentage of participants with clinically significant change from baseline in laboratory parameters. | week 0-26

CONTACTS AND LOCATIONS:
Locations (46):
- China (46):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The Second People's Hospital of Heifei, Hefei, Anhui
  - Ma'anshan People's Hospital, Ma’anshan, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Ninth People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - The First People's Hospital of Nanning, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Third People's Hospital of Hebei, Wuhan, Hubei
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Xuzhou Third People's Hospital, Xuzhou, Jiangsu
  - Nanchang First Hospital, Nanchang, Jiangxi
  - Affiliated Hospital of Changchun University of Chinese Medicine, Changchun, Jilin
  - Jilin Province FAW General Hospital, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Meihekou Central Hospital, Tonghua, Jilin
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liangning
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Jinan Central Hospital, Jinan, Shandong
  - Weifang Traditional Chinese Hospital, Weifang, Shandong
  - Shanghai Pudong Hospital, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Peace Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Jincheng General Hospital, Jincheng, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of The Fourth Military Medical University, Xian, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University (Xibei Hospital), Xian, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong Univesity, Xi’an, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang